CLINICAL TRIAL: NCT01254136
Title: A Phase I/II Study to Assess the Safety and Therapeutic Effect of INCB007839 in Combination With Trastuzumab and Vinorelbine in Patients With Metastatic HER2+ Breast Cancer.
Brief Title: Safety and Efficacy of INCB007839 With Trastuzumab and Vinorelbine in Patients With Metastatic HER2+ Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Incyte has suspended development of the compound.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 7839-204
Record Dates: First submitted 2010-12-01; First posted 2010-12-06 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — BID protein, human; Trastuzumab; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment A - INCB007839 300mg BID (Experimental): This is a single arm, open label study in which all patients will receive a single dose of the investigational product INCB007839 in combination with a standard regimen of trastuzumab and vinorelbine.
  Interventions: Drug: INCB007839 300mg BID; Drug: Trastuzumab; Drug: Vinorelbine

INTERVENTIONS:
Drug: INCB007839 300mg BID — INCB007839 tablets (300 mg BID) in combination with trastuzumab and vinorelbine will be administered in an initial Cycle of 28 days and followed by continuous 21-day cycles subsequently. Trastuzumab will be administered in continuous 21-day cycles beginning on Day 8 of Cycle 1. Vinorelbine will be administered on a weekly schedule for a minimum of the first four cycles beginning on Cycle 1 Day 8. All drugs will be administered continuously as tolerated or until a protocol-defined stopping criteria is met.
Drug: Trastuzumab — INCB007839 tablets (300 mg BID) in combination with trastuzumab and vinorelbine will be administered in an initial Cycle of 28 days and followed by continuous 21-day cycles subsequently. Trastuzumab will be administered in continuous 21-day cycles beginning on Day 8 of Cycle 1. Vinorelbine will be administered on a weekly schedule for a minimum of the first four cycles beginning on Cycle 1 Day 8. All drugs will be administered continuously as tolerated or until a protocol-defined stopping criteria is met.
Drug: Vinorelbine — INCB007839 tablets (300 mg BID) in combination with trastuzumab and vinorelbine will be administered in an initial Cycle of 28 days and followed by continuous 21-day cycles subsequently. Trastuzumab will be administered in continuous 21-day cycles beginning on Day 8 of Cycle 1. Vinorelbine will be administered on a weekly schedule for a minimum of the first four cycles beginning on Cycle 1 Day 8. All drugs will be administered continuously as tolerated or until a protocol-defined stopping criteria is met.

SUMMARY:
This Phase I/II study is designed to assess the safety and therapeutic effect of INCB007839 in combination with trastuzumab and vinorelbine in patients with metastatic HER2+ breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subject with diagnosis of metastatic (or locally recurrent-inoperable) breast cancer
* Subject with histological HER2+ status as determined by FISH with a gene amplification score of ≥ 2.2
* Subject with availability of archival biopsy tissue from primary tumor or metastatic lesions
* Subject with presence of measurable disease based on RECIST 1.1
* Subject who has received no more than three prior HER2-directed therapeutic regimens for advanced breast cancer

Exclusion Criteria:

* Subject with Left ventricular ejection fraction (LVEF) below institutional normal range
* Subject with metastasis to the central nervous system UNLESS asymptomatic and clinically stable
* Subject with current active malignancy other than breast cancer
* Subject with prior history of other malignancy except for cancers from which the patient is currently disease free
* Subject with significant renal or hepatic dysfunction
* Subject with history of venous or arterial thrombosis or risk factor for thrombosis other than history of malignancy
* Subject with insufficient bone marrow function
* Subject with contraindication to vinorelbine, trastuzumab, aspirin and/or warfarin therapy.
* Subject with current active bacterial, Hepatitis B or C, and/or HIV infections

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety and tolerabilty as determined by monitoring the frequency and severity of adverse events (AEs) and performing clinical assessments and laboratory investigations. | Measured monthly starting at Baseline (estimated duration 6-9 months)

SECONDARY OUTCOMES:
Overall objective response rate assessed by RECIST criteria | Measured at Baseline, Cycle 4 and approximately every 9 weeks after (estimated duration 6-9 months)

CONTACTS AND LOCATIONS:
Overall Officials: Denise A. Yardley, MD, Principal Investigator — Sara Cannon Research Institute
Locations (14):
- United States (14):
  - Fayetteville, Arkansas
  - Duarte, California
  - Denver, Colorado
  - Davie, Florida
  - Jacksonville, Florida
  - Detroit, Michigan
  - St Louis, Missouri
  - Hackensack, New Jersey
  - Lake Success, New York
  - Huntersville, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Salt Lake City, Utah